CLINICAL TRIAL: NCT01934062
Title: Induction Hypotension in Pediatric Population
Status: Completed | Type: Observational
Sponsor: Tariq Wani (Other)
Responsible Party: Sponsor-Investigator, Tariq Wani, Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00508
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Pediatric Surgical Patients
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical patients: Pediatric patients having surgery at Nationwide Children's Hosp. between 1/1/2013 & 7/31/2013.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — All surgeries performed at Nationwide Children's Hosp. between 1/1/2013 & 7/31/2013.
  --------------------------------------------------------------------------------

SUMMARY:
This is a retrospective chart review to assess the incidence and the degree of blood pressure changes after induction of anesthesia and to study the effect of different induction agents on blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients between ages of 1 year to 8 years will be included in the study.
* Patients with ASA physical classification 1 and 2 will be studied.

Exclusion Criteria:

* Patients with any cardiovascular or kidney diseases will be excluded from the study.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Surgical patients from Nationwide Children's Hosp.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Hypotension | Baseline, 5, 10, & 15 mins. post induction
  Measure the degree of change from pre-induction levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States